CLINICAL TRIAL: NCT04343599
Title: Hypopressive Effectiveness in Postural Control and Pelvic Floor.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, DAVID CRUZ DÍAZ, Professor, University of Jaén
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: Hypouja
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2020-04-13 (Actual); Status verified 2020-04

CONDITIONS: Pelvic Floor Disorders; Postural; Defect; Muscle Weakness
MeSH Terms: conditions — Pelvic Floor Disorders; Muscle Weakness

STUDY DESIGN:
Intervention Model Description: This study was a single-blinded randomized controlled trial
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: An independent assessor blinded to the data collection was responsible for the allocation process. A list of the computer-generated number was employed to assign participants to experimental or control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypopressive exercises (Experimental): Patients completed 10 weeks of abdominal hypopressive exercises with two sessions of 30 minutes per week.
  Interventions: Other: Hypopressive exercises
- Control group (No Intervention): Patients allocated to the control group did not receive any treatment.

INTERVENTIONS:
Other: Hypopressive exercises — The first two sessions will have as objective the correct and effective learning of the hypopressive technique. The rest of the sessions will be dedicated to the realization of an exercise protocol based on a progression of postures from standing to supine. Diaphragmatic apneas of approximately 7 seconds will be performed, alternating each apnea with three breaths.
  Arms: Hypopressive exercises

SUMMARY:
Effects of an exercise program based on hypopressive exercises in the female population.

DETAILED DESCRIPTION:
Participants allocated to the intervention group completed 10 weeks of hypopressive exercises training with a frequency of two sessions of 30 minutes twice a week.

ELIGIBILITY:
Inclusion Criteria:

* Women
* Physical autonomy

Exclusion Criteria:

* Vestibular disorders.
* Coronary diseases.
* Recent surgery.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-06-07 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Postural control | From baseline to 10 weeks.
  Postural control was evaluated by means of a stabilometric platform of resistive pressure sensors (Sensor Medica, Rome, Italy).

SECONDARY OUTCOMES:
Pelvic floor muscles strength | From baseline to 10 weeks.
  The assessment of the overall contractility of the striated pelvic floor musculature was evaluated according to the modified manual scale Oxford.
Self-reported pelvic floor status | From baseline to 10 weeks
  To assess self-reported status the Pelvic Floor Distress Inventory-Short Form was administered.
Urinary incontinence | From baseline to 10 weeks
  To determine the presence and improvement in urinary incontinence the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form was employed.
Transversus abdominis activation | From baseline to 10 weeks.
  Transversus abdominis thickness during contraction was assessed by real time ultrasound imaging.
Pulmonary ventilation | From baseline to 10 weeks
  A forced spirometry test was employed to assess pulmonary function.

CONTACTS AND LOCATIONS:
Overall Officials: David Cruz-Díaz, Principal Investigator — University of Jaén
Locations (1):
- University of Jaen, Jaén, Spain

IPD SHARING:
Plan to Share IPD: No
Provided by reasonable request.